CLINICAL TRIAL: NCT04135326
Title: Transcranial Direct Current Stimulation (tDCS) to Reduce Pain in Patients With Chemotherapy Induced Peripheral Neuropathy: A Pilot Study
Brief Title: Transcranial Direct Current Stimulation in Reducing Pain in Cancer Patients With Chemotherapy Induced Peripheral Neuropathy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Per PI termination request, no patients enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0541; NCI-2019-03834 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0541 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-10-10; First posted 2019-10-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2020-11

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (tDCS) (Experimental): Patients undergo tDCS QD over 20 minutes 5 days each week (Monday-Friday) for 3 weeks.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Transcranial Direct Current Stimulation

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Transcranial Direct Current Stimulation — Undergo tDCS
  Other Names: tDCS

SUMMARY:
This early phase I trial studies how well transcranial direct current stimulation works in reducing pain in cancer patients with chemotherapy induced peripheral neuropathy. Transcranial direct current stimulation is used for patients with brain injuries such as strokes as well as for mental health issues such as depression and may help to control pain in cancer patients with chemotherapy induced peripheral neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of transcranial direct current stimulation (tDCS) in reducing chemotherapy induced painful peripheral neuropathy (CIPPN).

Ia. Evaluate the change in pain scores Ib. Assess for changes in other symptoms (i.e insomnia, feeling of well-being, depression and anxiety).

SECONDARY OBJECTIVES:

I. To evaluate the following with the treatment of tDCS:

Ia. Assess for changes in using pain medications. Ib. Assess for changes in functioning (daily activities). Ic. Assess for changes in quality of life. Id. Assess for changes in neuropathy. Ie. Assess overall satisfaction with the tDCS treatment.

TERTIARY OBJECTIVES:

I. To evaluate tDCS treatment related side-effects.

OUTLINE:

Patients undergo tDCS once daily (QD) over 20 minutes 5 days each week (Monday-Friday) for 3 weeks.

After completion of study treatment, patients are followed up weekly for 3 weeks and at 4-6 weeks.

ELIGIBILITY:
Inclusion:

* Age greater than or equal to 18 years.
* Able to give a Voluntary written consent.
* Cancer patients with chemotherapy induced peripheral neuropathy of at least 3 months duration..
* Pain and/or tingling of at least 4/10

Exclusion:

* History of seizure
* History of migraine headache
* History of brain cancer and/or brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Change in chemotherapy induced peripheral neuropathy pain score | Baseline up to final day of treatment (3 weeks)
  The Pain inventory is an assessment of pain level on a 11-point numeric rating scales (0=none to 10=worst).

SECONDARY OUTCOMES:
Change in total opioid requirement (morphine equivalent daily dosage) | Baseline up to 4-6 weeks post-treatment
  Will be summarized using descriptive statistics including mean, standard deviation, median, range, and CIs.
Change in cancer related symptoms | Baseline up to 4-6 weeks post-treatment
  We will analyze each patient's Pain Management Center Follow-Up/ Progress Notes and Standardize questionnaire which includes the assessment of the aforementioned symptoms on a 11-point numeric rating scales (0=none to 10=worst).
Change in functioning of Daily Activities | Baseline up to 4-6 weeks post-treatment
  We will analyze each patient's Pain Management Center Follow-Up/ Progress Notes and Standardize questionnaire which includes the assessment of the aforementioned symptoms on a 11-point numeric rating scales (0=none to 10=worst).
Change in quality of life questionnaire | Baseline up to 4-6 weeks post-treatment
  We will analyze each patient's Pain Management Center Follow-Up/ Progress Notes and Standardize questionnaire which includes the assessment of the aforementioned symptoms on a 11-point numeric rating scales (0=none to 10=worst).
Incidence of adverse events | Up to 4-6 weeks post-treatment
  Frequency counts and percentages will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Salahadin Abdi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT04135326/ICF_000.pdf